CLINICAL TRIAL: NCT00911430
Title: Host Factors in Invasive and Recurrent Staphylococcus Aureus Infection
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090157; 09-I-0157
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-09-17

CONDITIONS: Staphylococcal Aureus Infection; Recurrent Staphylococcal Infection; Invasive Staphylococcal Infection
Keywords: Staphylococcus Aureus (S. Areus); Recurrent Staphylococcal Infection; Atopic Dermatitis; Immunodeficiency; Community Associated Staphylococcal Infection; Staphylococcal Infection; Invasive Staphylococcal Infection; Staph Infection
MeSH Terms: conditions — Staphylococcal Infections; Dermatitis, Atopic; Immunologic Deficiency Syndromes

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The incidence of community-associated (CA) staphylococcal infections, especially those caused by methicillin-resistant Staphylococcus aureus (MRSA), has increased dramatically in recent years. Although the majority of these infections are limited to the skin and soft tissue and thus not life threatening, the number of invasive cases in otherwise healthy individuals is increasing and some are fatal. As a first step toward understanding pathogenesis, there has been significant focus on elucidating the key CA-MRSA virulence factors. The relative significance of these factors is still being delineated. By comparison, there has been little focus on host factors associated with these invasive infections. In this protocol, we will recruit 100 otherwise healthy subjects with invasive staphylococcal infection, 50 otherwise healthy subjects with recurrent staphylococcal infections, and obtain samples from 150 unidentified healthy controls from the blood bank to investigate host immunologic factors predisposing people to staphylococcal infection. Subjects will receive standard of care treatment for acute or recurrent staphylococcal infections. The primary objective of this research is to identify host genetic factors that contribute to susceptibility or severity of community acquired staphylococcal diseases. We will use three experimental approaches to complete this objective: 1) expression microarray analyses of study population s (subjects and controls) white cells (neutrophils and peripheral blood mononuclear cells) at rest and stimulated with staphylococci, 2) evaluation of toll-like receptor (TLR) pathways in the study population s cells, and 3) evaluation of Th17 cells. The proposed research will address a key area of staphylococcal pathogenesis for which there is a striking lack of information. We fully anticipate that the research also will provide critical new information directly relevant to vaccine, diagnostics, and therapeutics development.

DETAILED DESCRIPTION:
The incidence of community-associated (CA) staphylococcal infections, especially those caused by methicillin-resistant Staphylococcus aureus (MRSA), has increased dramatically in recent years. Although the majority of these infections are limited to the skin and soft tissue and thus not life threatening, the number of invasive cases in otherwise healthy individuals is increasing and some are fatal. As a first step toward understanding pathogenesis, there has been significant focus on elucidating the key CA-MRSA virulence factors. The relative significance of these factors is still being delineated. By comparison, there has been little focus on host factors associated with these invasive infections. In this protocol, we will recruit 100 otherwise healthy subjects with invasive staphylococcal infection, 50 otherwise healthy subjects with recurrent staphylococcal infections, and obtain samples from 150 unidentified healthy controls from the blood bank to investigate host immunologic factors predisposing people to staphylococcal infection. Subjects will receive standard of care treatment for acute or recurrent staphylococcal infections. The primary objective of this research is to identify host genetic factors that contribute to susceptibility or severity of community acquired staphylococcal diseases. We will use three experimental approaches to complete this objective: 1) expression microarray analyses of study population s (subjects and controls) white cells (neutrophils and peripheral blood mononuclear cells) at rest and stimulated with staphylococci, 2) evaluation of toll-like receptor (TLR) pathways in the study population s cells, and 3) evaluation of Th17 cells. The proposed research will address a key area of staphylococcal pathogenesis for which there is a striking lack of information. We fully anticipate that the research also will provide critical new information directly relevant to vaccine, diagnostics, and therapeutics development.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age greater than or equal to 2 years.
  2. Current or past S. aureus infection, either invasive or soft tissue.
  3. Willingness to allow storage of blood and tissue samples for future use.
  4. Subjects will be eligible without regard to race, gender, or ethnic origin.

EXCLUSION CRITERIA:

1. Infection with known HIV-1, HIV-2 as demonstrated by ELISA and Western blot or viral load testing.
2. Evidence of intravenous drug abuse in the year prior to the first (or only) S. aureus infection.
3. Previously known immunodeficiency syndrome.
4. Evidence of active malignancy.
5. Any condition that the investigators judge would compromise the results of the study.
6. Diabetes mellitus.
7. Evidence of healthcare-associated infection invasive device, history of surgery with implantation of artificial device in previous 12 months, history of surgery without device implantation in previous 12 month, or dialysis, hospitalization, or residence in long-term care facility in previous 12 months. An exception to these exclusion criteria is hospitalization for the acute S. aureus infection at the time of enrollment.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-05-28; Study Completion 2014-09-17

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Holland, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Diekema DJ, Pfaller MA, Schmitz FJ, Smayevsky J, Bell J, Jones RN, Beach M; SENTRY Partcipants Group. Survey of infections due to Staphylococcus species: frequency of occurrence and antimicrobial susceptibility of isolates collected in the United States, Canada, Latin America, Europe, and the Western Pacific region for the SENTRY Antimicrobial Surveillance Program, 1997-1999. Clin Infect Dis. 2001 May 15;32 Suppl 2:S114-32. doi: 10.1086/320184. PMID 11320452
- [Background] Zetola N, Francis JS, Nuermberger EL, Bishai WR. Community-acquired meticillin-resistant Staphylococcus aureus: an emerging threat. Lancet Infect Dis. 2005 May;5(5):275-86. doi: 10.1016/S1473-3099(05)70112-2. PMID 15854883
- [Background] Naimi TS, LeDell KH, Como-Sabetti K, Borchardt SM, Boxrud DJ, Etienne J, Johnson SK, Vandenesch F, Fridkin S, O'Boyle C, Danila RN, Lynfield R. Comparison of community- and health care-associated methicillin-resistant Staphylococcus aureus infection. JAMA. 2003 Dec 10;290(22):2976-84. doi: 10.1001/jama.290.22.2976. PMID 14665659